CLINICAL TRIAL: NCT05385887
Title: Antibiotic Treatment foLlowing Surgical drAinage of Perianal abScess; the ATLAS Trial, a Double-blind, Placebo-controlled, Randomized Trial
Brief Title: Antibiotic Treatment foLlowing Surgical drAinage of Perianal abScess; the ATLAS Trial
Acronym: ATLAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: dr. IJM Han-Geurts (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor-Investigator, dr. IJM Han-Geurts, Principal investigator, Proctos Kliniek
Organization: Proctos Kliniek (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL75540.018.20; 2020-004449-35 (EudraCT Number)
Record Dates: First submitted 2022-05-12; First posted 2022-05-23 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Perianal Fistula; Perianal Abscess; Drain Abscess
Keywords: antibiotics; antibiotic treatment; perianal fistula; perianal abscess; drainage of abscess
MeSH Terms: interventions — Ciprofloxacin; Metronidazole

STUDY DESIGN:
Intervention Model Description: double-blind, placebo-controlled, randomized trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patiënt, clinician and investigators are all blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antibiotic treatment (Active Comparator): Two kinds of antibiotics: Ciprofloxacine 500mg 2dd & Metronidazole 500mg 3dd
  Interventions: Drug: Ciprofloxacin 500 mg; Drug: Metronidazole 500 mg
- Placebo (Placebo Comparator): Placebo tabletes
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciprofloxacin 500 mg — One tablet of 500mg Ciprifloxacine, twice a day
  Arms: Antibiotic treatment
Drug: Metronidazole 500 mg — One tablet of 500mg Metronidazole, three times a day
  Arms: Antibiotic treatment
Drug: Placebo — Placebo tablets
  Arms: Placebo

SUMMARY:
Rationale:

Perianal fistula is a burdening disease with an annual prevalence of 2/100.000 in the Dutch population. More than 90% of crypto-glandular fistulas originate from anorectal abscess. Despite adequate drainage of anorectal abscess up to 83% recurs or results in an anal fistula, the majority developing within 12 months. Up till now it is not common practice to routinely administer prophylactic antibiotics to prevent anal fistula development.\

Objective:

The objective of this trial is to establish if adding antibiotic treatment to surgical drainage of perianal abscess results in less perianal fistulas.

Study design:

The study concerns a double-blind, placebo-controlled, randomized, multicenter trial with treatment of perianal abscess by surgical drainage alone or combined with antibiotic treatment. Patients will be accrued by all participating clinics. The design involves allocation of all appropriate consecutive patients with a primary occurrence of perianal abscess to surgical drainage followed by either antibiotics or placebo. Data will be analyzed on 'intention to treat' basis in case patients are not subjected to the randomized treatment modality.

Study population:

Men and women of 18 years and older who present for the first time with a perianal abscess.

Intervention (if applicable): The antibiotic group receives 7 days of oral metronidazole (500 mg every eight hours) and ciprofloxacin (500 mg every twelve hours) in addition to surgical drainage. The other group receives surgical drainage and postoperatively identical placebo tablets.

Main study parameters/endpoints:

Primary outcome measure is development of a perianal fistula. Secondary outcome measures are quality of life at 12 months measured with the EQ-5D-5L with Dutch rating. Further: in-hospital direct and indirect costs and out-of hospital postoperative costs, need of repeated drainage, patient related outcome (PRO) and clinical outcome measures.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

For this study, patients are asked to take part in a study comparing the addition of antibiotic treatment to surgical drainage of perianal abscess. Patients will not be burdened by extra hospital visits. At baseline participants will complete PRO questionnaires. Also at 1 week and 3, 6 and 12 months participants will fulfill the PRO questionnaires. These will be send to them by email and will take approximately 10 minutes each time.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years or older
* Eligible for e-mail questionnaires
* Sufficient understanding of the Dutch written language (reading and writing)
* Obtained written informed consent

Exclusion Criteria:

* A coexistent anorectal fistula
* Secondary or recurrent anorectal abscess
* Presence of an internal fistula opening
* Any additional surgical procedure performed during the same session
* Previous (peri)anal surgery
* Inflammatory bowel disease
* History of radiation of the pelvic area
* Anorectal malignancy
* Immunodeficiency
* Kidney failure (eGFR <30ml/min)
* Valvular heart disease
* Pregnancy or lactation
* Postoperative antibiotic prophylaxis indicated for another reason
* Immunosuppressive medication at the time of surgery
* Allergy to metronidazole or ciprofloxacin
* Not able or trouble with swallowing pills
* Concomitant use of:

  * Tizanidine, theophylline, clozapine, olanzapine, pirfenidone, carbamazepine, agomelatine (these are all CYP1A2 substrates, ciprofloxacin is an inhibitor)
  * Amiodarone, erythromycin, sotalol, azithromycin, citalopram, escitalopram, flecainide, fluconazole, haloperidol >5mg/day, methadone, ondansetron (concerning prolonged QT interval in combination with ciprofloxacin)
  * Lithium (can cause toxic levels with metronidazole)
  * Lopinavir/ritonavir, ritonavir capsules, temsirolimus, disulfiram (antabuse), mebendazole (can cause serious side effects, confusion and psychosis in combination with metronidazole)
  * Corticosteroids (in combination with ciprofloxacin higher risk of tendinitis and tendon rupture).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Estimated)
Dates: Start 2021-12-23 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Perianal fistula at 1 year follow up | 1 year
  A perianal fistula is diagnosed based on findings from physical examination or by a telephone call after 12 months were the doctor asks for symptoms as serosanguinous discharge and pain. An external opening with or without serosanguilent discharge is considered a fistula. In case of doubt an endoanal ultrasonography or MRI is performed.
  So: yes/no fistula (dichotomous parameter)

SECONDARY OUTCOMES:
Quality of life at 12 months measured with the EQ-5D-5L with Dutch rating. | 1 year
  The EQ-5D-5L is a generic Health Related Quality of Life (HRQoL) measure, which is broadly used in economic evaluation. The instrument examines a patient's HRQoL on the day of the interview. It consists of the EQ-5D-5L descriptive system and the EQ-Visual Analogue Scale. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has five levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Responses to the 5 items result in a patient's health state that can be transformed into an index score representing health-related quality of life, ranging between 0 (death) and 1 (full health). These index scores are combined with length of life to calculate the QALY. The EQ-VAS records the patient's self-rated health with endpoints labelled 'the best health you can imagine' at the top and 'the worst health you can imagine' at the bottom.
In-hospital direct and indirect costs and out-of hospital posteroperative costs | 1 year
  In-hospital direct and indirect costs (measured with iPCQ and iMCQ) and out-of hospital postoperative costs.
Need of repeated drainage | 1 year
PROMs | 1 year
  Patient related outcome (PRO) are complaint reduction assessed by a proctology specific validated patient-related outcome measure, the proctoPROM(14). This was recently developed and validated at Proctos Clinic. At baseline participants will complete PRO questionnaires. Also at 1 week and 3, 6 and 12 months participants will fulfill the PRO questionnaires. These will be send to them by email with access to a web tool (Castor). If the patient does not have an email account, the questionnaires will be send the patients' home address, accompanied by a return envelope provided with postage stamps and the address of the hospital.
Day of discharge from hospital | 1 year
  Day of discharge from hospital;
Postoperative complications | 1 year
  Complications (postoperative bleeding, urinary retention requiring catheterisation, emergency reoperation, anal stenosis and fecal incontinence) including death and cause of death within 30 days will be reported using the Clavien-Dindo classification of surgical complications(15).
Recurrent abscess | 1 year
  (Recurrent) abscess within one year. Yes/no (dichotomous)
Duration of absence from work | 1 year
  Duration of absence from work. Amound of days is recorded (continuous scale)

CONTACTS AND LOCATIONS:
Locations (11):
- Netherlands (11):
  - Amphia hospital, Breda, North Brabant
  - Elisabeth-TweeSteden ziekenhuis, Tilburg, North Brabant
  - OLVG, Amsterdam, North Holland
  - Rode Kruis ziekenhuis, Beverwijk, North Holland
  - Dijklander hospital, Hoorn, North Holland
  - Albert Schweitzer ziekenhuis, Dordrecht, South Holland
  - Proctos kliniek, Bilthoven, Utrecht
  - Flevoziekenhuis, Almere Stad
  - University Medical Center location AMC, Amsterdam
  - IJsselland ziekenhuis, Capelle aan den IJssel
  - Diakonessenhuis, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
A data management plan (DMP) will be composed containing the FAIR principles. Existing data will be used, and new data will be generated. Data are registered in an archive or repository and open access will be enabled. Results will be disclosed in a peer review medical journal to guarantee transparency. The study protocol was registered in an open access public trial registry before recruitment started.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within one year after the last study visit of the last patient. Data will be availabe for 15 years.

REFERENCES:
- [Derived] van Oostendorp JY, Dekker L, van Dieren S, Bemelman WA, Han-Geurts IJM. Antibiotic Treatment foLlowing surgical drAinage of perianal abScess (ATLAS): protocol for a multicentre, double-blind, placebo-controlled, randomised trial. BMJ Open. 2022 Nov 8;12(11):e067970. doi: 10.1136/bmjopen-2022-067970. PMID 36351727